CLINICAL TRIAL: NCT06161948
Title: The Effect of Time-restricted Enteral Nutrition on the Prognosis of Severe Stroke Patients: a Multicentre, Prospective, Randomised, Open-label, Blinded-endpoint Trial
Brief Title: Time-restricted Enteral Nutrition Versus Continuous Enteral Nutrition in Patients With Severe Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023AH040243
Record Dates: First submitted 2023-11-19; First posted 2023-12-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Time Restricted Feeding
MeSH Terms: conditions — Stroke; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted group (Experimental): Time-restricted enteral nutrition therapy group
  Interventions: Other: Time-restricted enteral nutrition therapy group
- Continuous group (Other): Continuous enteral nutrition control group
  Interventions: Other: Continuous enteral nutrition control group

INTERVENTIONS:
Other: Time-restricted enteral nutrition therapy group — Control the daily enteral nutrition time to 8-12 hours, enteral nutrition start time: 06:00 ~ 08:00, end time: 16:00 ~ 18:00. Enteral nutrition lasts until the patient discontinues enteral nutrition, the patient dies, the patient is transferred from the ICU, or enteral nutrition is used until 28 days, whichever event occurs first.
  Arms: Time-restricted group
Other: Continuous enteral nutrition control group — The control group was continuous enteral nutrition (24 hours), which lasted until the patient stopped taking enteral nutrition, the patient died, the patient was transferred from the ICU, or enteral nutrition was used until 28 days, whichever event occurred first.
  Arms: Continuous group

SUMMARY:
In patients with severe stroke whose GCS score is ≤12 points or NIHSS score is ≥11 points, to evaluate whether time-restricted enteral nutrition can improve the incidence of poor 90-day prognosis (mRS ≥3 points) compared with continuous enteral nutrition.

DETAILED DESCRIPTION:
Control the daily enteral nutrition time to 8-12 hours, enteral nutrition start time: 06:00 ~ 08:00, end time: 16:00 ~ 18:00. Enteral nutrition lasts until the patient discontinues enteral nutrition, the patient dies, the patient is transferred from the ICU, or enteral nutrition is used until 28 days, whichever event occurs first.

On the first day of enrollment: the patient is given 1/3 of the estimated energy and 1.2-1.5g/kg/d of protein through enteral nutrition; On the second day of enrollment: the patient is given 1/2 of the estimated energy and 1.2-1.5g/kg/d of protein through enteral nutrition; Enrollment 3 - End of intervention: The patient is given 100% of the estimated energy through enteral nutrition, which can fluctuate between 70% and 100% of the estimated energy, and the protein is 1.2-1.5g/kg/d.

The control group was continuous enteral nutrition (24 hours), which lasted until the patient stopped taking enteral nutrition, the patient died, the patient was transferred from the ICU, or enteral nutrition was used until 28 days, whichever event occurred first.

On the first day of enrollment: the patient is given 1/3 of the estimated energy and 1.2-1.5g/kg/d of protein through enteral nutrition; On the second day of enrollment: the patient is given 1/2 of the estimated energy and 1.2-1.5g/kg/d of protein through enteral nutrition; Enrollment 3 - End of intervention: The patient is given 100% of the estimated energy through enteral nutrition, which can fluctuate between 70% and 100% of the estimated energy, and the protein is 1.2-1.5g/kg/d.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and <80 years old;
* Cerebral parenchymal hemorrhage or cerebral infarction within 72 hours of onset;
* GCS score ≤12 points or NIHSS score ≥11 points on admission,
* Enteral nutrition is planned, and the estimated enteral nutrition treatment time is ≥7 days;
* Signed informed consent form.

Exclusion Criteria:

* Complete parenteral nutrition is required due to contraindications to enteral nutrition;
* After gastrectomy or intestinal resection;
* Enteral nutrition treatment has been performed for >12 hours;
* Accompanying diseases: a. Advanced cancer; b. Severe cardiac insufficiency [ejection fraction ≤ 50%]; c. Severe liver failure [Child Pugh score ≥ 7]; d. Severe renal failure [glomerular filtration] rate ≤ 30 mL/min or serum creatinine ≥ 4 mg/dL])
* Have a history of mental illness or mRS ≥ 3 points;
* The patient's doctor or nutritional therapist believes that the plan is not in the best interest of the patient;
* During the patient's admission, death is inevitable, and there are underlying diseases that result in a survival time of <90 days;
* The patient participates in another clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Poor 90-day functional prognosis | Day 90 post-randomization
  mRS ≥ 3 points

SECONDARY OUTCOMES:
GCS score at discharge | The day of Discharge, an average of 20 days
  Glasgow Coma Scale,the score ranges from 3-15. The lower the score, the greater the impairment of consciousness
NIHSS score at discharge | The day of Discharge, an average of 20 days
  NIH Stroke Scale,the score ranges from 0~42 points, and the higher the score, the more severe the nerve damage
mRS score at discharge | The day of Discharge, an average of 20 days
  Modified Rankin Scale，the score ranges from 0~6 levels,and the higher the score, the more severe outcome
Barthel index at discharge | The day of Discharge, an average of 20 days
  Barthel index at discharge
90-day Barthel Index | Day 90 post-randomization
  90-day Barthel Index
ICU length of stay | From admission to ICU to transfer out of ICU .an average of 11 days
  ICU length of stay
Length of hospital stay | The day of Discharge, an average of 20 days
  total length of stay

OTHER OUTCOMES:
Adverse events during hospitalization | From enrollment to discharge, an average of 20 days
  Safety outcomes
Serious adverse events during hospitalization | From enrollment to discharge, an average of 20 days
  Safety outcome
28-day mortality rate | From enrollment to Day 28 post-randomization
  Safety outcome
90-day mortality rate. | From enrollment to Day 90 post-randomization
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yu, doctor, Principal Investigator — First Affiliated Hospital of Wannan Medical College
Locations (1):
- The first affliated hospital of Wannan medical college, Wuhu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu T, Shi G, Ye Z, Jiang X, Jia W, Wang Y, Wang Y, Xu J. Rationale and design of a PROBE trial comparing continuous enteral nutrition to time-restricted enteral nutrition in severe stroke. Stroke Vasc Neurol. 2025 Dec 3:svn-2025-004382. doi: 10.1136/svn-2025-004382. Online ahead of print. PMID 41339081